CLINICAL TRIAL: NCT07329036
Title: The Artificial Liver Support System (ALSS) in Patients With Acute on Chronic Liver Failure - the Use of Combined Molecular Adsorption System With Double Plasma (DPMAS) and Therapeutic Plasma Exchange (TPE), Its Effect on Primary Coagulation and the Function of Vital Organs.
Brief Title: ALSS - DPMAS and Therapeutic Plasma Exchange (TPE), Its Effect on Primary Coagulation, Inflammation and the Function of Vital Organs in ALF or ACLF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Responsible Party: Principal Investigator, Petr Piza, anesthesiologist/intensivist, Institute for Clinical and Experimental Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Study1
Record Dates: First submitted 2024-02-29; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Acute Liver Failure
Keywords: acute liver failure
MeSH Terms: conditions — Liver Failure, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ALSS (alternating DPMAS and TPE) (Experimental): Participants meeting inclusion criteria will receive artificial liver support system (ALSS) therapy in addition to standard of care. ALSS sessions will be performed for up to 7-10 days or until liver transplantation or recovery of hepatic function, whichever occurs first. ALSS modalities will be alternated according to protocol (DPMAS and TPE alternating between sessions). Outcomes will be assessed through Day 28 after hospital admission (or per protocol).
  Interventions: Device: The artificial liver support system (ALSS) - DPMAS/TPE
- Standard care (No Intervention): Participants will receive standard of care for ACLF according to institutional protocol without ALSS (no DPMAS and no TPE as part of ALSS).

INTERVENTIONS:
Device: The artificial liver support system (ALSS) - DPMAS/TPE — Device: Double Plasma Molecular Adsorption System (DPMAS) Procedure/Other: Therapeutic Plasma Exchange (TPE)
  Arms: ALSS (alternating DPMAS and TPE)

SUMMARY:
The artificial liver support system (ALSS) in patients with acute on chronic liver failure - the use of combined molecular adsorption system with double plasma (DPMAS) and therapeutic plasma exchange (TPE), its effect on primary coagulation, inflammation and the function of vital organs.

DETAILED DESCRIPTION:
In patients with ACLF we assume the use of the proposed protocol of combined support therapy (consisting of a hemoadsorption system - DPMAS (double plasma molecular absorption system) and therapeutic plasma (TPE), with the basic aim of improving clinical condition (organ dysfunction) to allow the regeneration of liver parenchyma or to perform liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient, age ≥18 years
* Expressed consent to the inclusion
* Patient hospitalized on ICU with ALF or ACLF diagnosis
* Recently meeting the inclusion to liver transplantation
* Present on a waiting list to liver transplant
* Unsuitable for inclusion to liver transplantation - indicated for support therapy only, but not indented to palliative care

Exclusion Criteria:

* Disagreement with the study
* Infaust prognosis with expected survival less than 24 hours
* Physiologically/biologically very advanced stage patients condition, severe lung disease (Gold criteria 3 or 4), heart failure (functional class NYHA III or IV) or neurological disease, as well as ACLF-3.
* Advanced oncological disease (expected life expectancy below 6 months)
* Severe degree of Frailty syndrome in secondary severe sarcopenia (muscle and malnutrition) or reduced performance state according

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Transplant-Free Survival at Day 21 | 21 days after the first ALSS (DPMAS/TPE) session
  Proportion of patients with acute liver failure who are alive without liver transplantation at Day 21 after initiation of artificial liver support therapy (combined DPMAS + TPE).

SECONDARY OUTCOMES:
Overall Survival at Day 21 | 21 days after the first ALSS session
  Proportion of patients who are alive (with or without liver transplantation) at Day 21 after initiation of ALSS therapy.
Overall Survival at Day 90 | 90 days after the first ALSS session
  Proportion of patients who are alive (with or without liver transplantation) at Day 90 after initiation of ALSS therapy.
Liver Transplantation Rate and Timing | Up to 90 days after the first ALSS session
  Proportion of patients who undergo liver transplantation after initiation of ALSS therapy and time from ALSS initiation to liver transplantation (days).

OTHER OUTCOMES:
Change in Hepatic Encephalopathy Grade | Baseline (before first ALSS session) Daily for 7 days after ALSS initiation Day 14 Day 21
  West Haven grade (0-4)
Change in Plasma Ammonia Concentration | Baseline (within 6 hours before first ALSS session) Immediately after each ALSS session 24 hours after the final ALSS session Day 3, Day 7, Day 14, Day 21
  µmol/L
Change in International Normalized Ratio (INR) | Baseline: Within 1 hour before the first DPMAS + TPE session Immediate Post-Procedure: Within 1 hour after each ALSS session Early Post-Intervention: 24 hours after the final ALSS session Follow-Up: Day 3 and Day 7
  Unit of Measure: INR units
Change in C-reactive Protein (CRP) Concentration | Baseline 24 hours after each ALSS session 72 hours after the final ALSS session Day 7 Day 14
  mg/L
Change in Global Liver Disease Severity (Model for End-Stage Liver Disease [MELD] Score) | Baseline; Day 3; Day 7; Day 14; Day 21
  Change from baseline in the Model for End-Stage Liver Disease (MELD) score, a validated severity scale of chronic liver disease. The MELD score is calculated from serum bilirubin, serum creatinine, and INR (International Normalized Ratio). Score range: 6 to 40, with higher scores indicating more severe liver disease and worse prognosis. Change from baseline will be calculated at each time point as: (MELD at time point - MELD at baseline). MELD will be calculated using the standard formula.
Change From Baseline in Vasopressor Dose (Norepinephrine Equivalent Dose, NED) | Baseline; 24 hours after each ALSS session; daily until Day 7 (unit: µg/kg/min (norepinephrine equivalent))
  Norepinephrine equivalent dose (NED) will be recorded at baseline, 24 hours after each ALSS session, and then daily through Day 7. Change from baseline will be calculated at each time point as: (NED at time point - NED at baseline).
Incidence of Treatment-Emergent Adverse Events Related to ALSS (Combined DPMAS + TPE) | During each ALSS session; up to 7 days after the final ALSS session
  Number of participants with treatment-emergent adverse events (TEAEs) considered related to ALSS (combined DPMAS + TPE) occurring during each ALSS session or within 7 days after the final ALSS session, including: procedure-related bleeding, hemodynamic instability during the procedure, allergic or anaphylactic reactions, circuit clotting, and clinically significant electrolyte disturbances requiring intervention. Relationship to ALSS will be assessed by the investigator according to predefined criteria.
Change in Fibrinogen Concentration | Baseline: Within 1 hour before first DPMAS + TPE session Immediate Post-Procedure: Within 1 hour after each ALSS session Early Post-Intervention: 24 hours after the final ALSS session Follow-Up: Day 3 and Day 7
  Unit of Measure: g/L
Change in Platelet Count | Baseline: Within 1 hour before first DPMAS + TPE session Post-Procedure: Within 12 hour after each ALSS session Early Post-Intervention: 24 hours after the final ALSS session Follow-Up: Day 3 and Day 7
  Unit of Measure: ×10⁹/L
Change in Viscoelastic Clotting Time (ROTEM/TEG | Baseline: Within 1 hour before first DPMAS + TPE session Post-Procedure: Within 2 hour after each ALSS session Early Post-Intervention: 24 hours after the final ALSS session Follow-Up: Day 3 and Day 7
  Unit of Measure: Seconds
Change in Maximum Clot Firmness (ROTEM/TEG) | Baseline: Within 1 hour before first DPMAS + TPE session Post-Procedure: Within 2 hour after each ALSS session Early Post-Intervention: 24 hours after the final ALSS session Follow-Up: Day 3 and Day 7
  Unit of Measure: mm
Change in D-dimer Concentration | Baseline: Within 1 hour before first DPMAS + TPE session Immediate Post-Procedure: Within 12 hour after each ALSS session Early Post-Intervention: 24 hours after the final ALSS session Follow-Up: Day 3 and Day 7
  Unit of Measure: mg/L FEU
Change in Coagulation Factor VIII Activity | Baseline: Within 1 hour before first DPMAS + TPE session Immediate Post-Procedure: Within 1 hour after each ALSS session Early Post-Intervention: 24 hours after the final ALSS session Follow-Up: Day 3 and Day 7
  Unit of Measure: % activity
Change in von Willebrand Factor Antigen (vWF:Ag) | Baseline: Within 1 hour before first DPMAS + TPE session Immediate Post-Procedure: Within 1 hour after each ALSS session Early Post-Intervention: 24 hours after the final ALSS session Follow-Up: Day 3 and Day 7
  Unit of Measure: %
Change in von Willebrand Factor Activity (vWF:RCo or vWF:GPIbM) | Baseline: Within 1 hour before first DPMAS + TPE session Immediate Post-Procedure: Within 1 hour after each ALSS session Early Post-Intervention: 24 hours after the final ALSS session Follow-Up: Day 3 and Day 7
  Unit of Measure: %
Change in ADAMTS-13 Activity | Baseline: Within 1 hour before first DPMAS + TPE session Immediate Post-Procedure: Within 1 hour after each ALSS session Early Post-Intervention: 24 hours after the final ALSS session Follow-Up: Day 3 and Day 7
  Unit of Measure: % activity
Change in Protein C Activity | Baseline: Within 1 hour before first DPMAS + TPE session Immediate Post-Procedure: Within 1 hour after each ALSS session Early Post-Intervention: 24 hours after the final ALSS session Follow-Up: Day 3 and Day 7
  Unit of Measure: % activity
Change in Protein S Activity | Baseline: Within 1 hour before first DPMAS + TPE session Immediate Post-Procedure: Within 1 hour after each ALSS session Early Post-Intervention: 24 hours after the final ALSS session Follow-Up: Day 3 and Day 7
  Unit of Measure: % activity
Change in Procalcitonin (PCT) Concentration | Baseline 24 hours after each ALSS session 72 hours after the final ALSS session Day 7 Day 14
  ng/mL
Change in Interleukin-6 (IL-6) Concentration | Baseline 24 hours after each ALSS session 72 hours after the final ALSS session Day 7 Day 14
  pg/mL
Change in Total Serum Bilirubin | Baseline Daily for 7 days Day 14 Day 21
  µmol/L
Change in Alanine Aminotransferase (ALT) | Baseline Daily for 7 days Day 14 Day 21
  U/L
Change in Aspartate Aminotransferase (AST) | Baseline Daily for 7 days Day 14 Day 21
  U/L
Change in MELD Score (Model for End-Stage Liver Disease) | Baseline Day 3 Day 7 Day 14 Day 21
  Score on a scale from 6 to 40 Higher scores indicate worse liver disease severity.
Change from baseline in serum creatinine. | Baseline Daily for 7 days Day 14 Day 21
  µmol/L
Change in Blood Urea Nitrogen (BUN) | Baseline Daily for 7 days Day 14 Day 21
  mmol/L
Change in Urine Output | Baseline Daily for 7 days Day 14 Day 21
  mL/kg/hour
New requirement for renal replacement therapy compared with baseline. | Baseline Daily for 7 days Day 14 Day 21
  Yes/No
Change from baseline in vasopressor dose expressed as norepinephrine-equivalent rate. | Baseline (before first ALSS session) 24 hours after each ALSS session Daily through Day 7
  µg/kg/min
Change from baseline in mean arterial pressure | Baseline (before first ALSS session) 24 hours after each ALSS session Daily through Day 7
  mmHg
Change from baseline in the ratio of arterial oxygen partial pressure to inspired oxygen fraction. | Baseline Day 3 Day 7 Day 14
  Ratio (unitless)
New requirement for invasive mechanical ventilation compared with baseline | Baseline Day 3 Day 7 Day 14
  Yes/No
ICU Length of Stay | From ICU admission to ICU discharge, up to 28 days after ICU admission
  ICU length of stay is defined as the number of days from ICU admission (date/time) to ICU discharge (date/time).
Duration of Total Hospital Admission (Hospital Length of Stay) | From hospital admission to hospital discharge, up to 90 days after hospital admission
  Hospital length of stay is defined as the number of days from hospital admission (date/time) to hospital discharge (date/time).
Change From Baseline in Mean Arterial Pressure (MAP) | Baseline; 24 hours after each ALSS session; daily until Day 7 (unit: mmHg)
  Mean arterial pressure (MAP) will be recorded at baseline, 24 hours after each ALSS session, and then daily through Day 7. Change from baseline will be calculated at each time point as: (MAP at time point - MAP at baseline).

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Clinical and Experimental Medicine (IKEM), Prague, Czechia

IPD SHARING:
Plan to Share IPD: No